CLINICAL TRIAL: NCT05064852
Title: A Real-world Study of the Safety and Efficacy of Surufatinib in the Treatment of Biliary Tract Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: HMPL-012-RWS-BTC101
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surufatinib: Patients with BTC visited the site from 2021 to 2023 and received Surufatinib therapy.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — The study is a real-world study. According to the actual medical history of patients, the usage of Surufatinib was collected.

SUMMARY:
This is a prospective, single-arm, open-label,multi-center, observational real-world clinical study to observe and evaluate the efficacy and safety of Surufatinib in the treatment of patients with biliary tract cancer (BTC).

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label,multi-center, observational real-world clinical study to observe and evaluate the efficacy and safety of Surufatinib in the treatment of patients with biliary tract cancer (BTC). About 200 subjects are prepared to recruit in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male or female;
2. Patients with histologically or cytologically confirmed unresectable or metastatic BTC, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC), and gallbladder cancer (GBC); Surgical resection with positive margins are allowed;
3. ECOG score 0-2;
4. Expected survival of ≥12 weeks;
5. Confirmed measurable (or evaluable) lesions that meet the requirements of RECIST 1.1;
6. It is not less than 7 days since the end of the last systematic treatment, and the palliative treatment of the limited area is allowed

   Treatment has been over 4 weeks;
7. The function of major organs and bone marrow was basically normal;
8. Fully understand this study, voluntarily participate in it, and sign the informed consent.
9. Fertile male or female patients shall volunteer to use effective contraceptive methods, such as double barrier contraception, condoms, oral or injected contraceptives, and intrauterine devices, during the study period and within 90 days after the last dosing of the investigational drug. All-female patients will be considered fertile unless they have had natural menopause, or artificial menopause, or sterilization (such as hysterectomy, bilateral adnexectomy, or ovarian radiation)

Exclusion Criteria:

1. Fine basal skin that has been diagnosed with other malignant tumors within the past 5 years and has been effectively treated (Except for cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer and breast cancer after effective resection outside);
2. Receiving other investigational drugs or approved or under development antitumor therapies;
3. Patients with contraindications to Surufatinib (e.g., active bleeding, ulcers, intestinal perforation, bowel)Obstruction, medically uncontrolled hypertension, grade III-IV cardiac dysfunction, major surgery within 30 days, severe liver and kidney insufficiency, etc.);
4. The patient has any current disease or condition that affects the absorption of the drug, or the patient cannot take it orally Surufatinib;
5. Demonstrated allergy to any component of the test drug and/or its excipients;
6. Pregnant (positive pregnancy test before dosing) or breast-feeding women;
7. Patients with large pleural effusion or ascites requiring drainage;
8. Taken a drug containing hyperforin perforatum within 3 weeks prior to the first study, or before taken other CYP3A4 strong inducer or inhibitor within 2 weeks;
9. The investigator determined that liver metastases accounted for 50% or more of the total volume of the liver;
10. Clinically intervened biliary obstruction was not in remission or required anti-infective therapy as determined by the investigator 14 days prior to the first study drug treatment;
11. Previous liver transplantation;
12. Clinically significant electrolyte abnormalities as determined by the investigator;
13. Any other diseases with clinically significant metabolic abnormalities, abnormal physical observations, or abnormal laboratory findings, which are judged by the investigator as evidence that the patient has a disease or condition that is unsuitable for the study drug (e.g., epileptic seizures requiring treatment), or that would interfere with the interpretation of the study results, or that may put the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Biliary Tract Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months after the last patient enrolled
  PFS was defined as the length of time from the administration of the first-dose until disease progression or death from any cause before disease progression.

SECONDARY OUTCOMES:
Safty | up to 4 weeks after the last dose
  The rate of AE and SAE in patients with BTC receiving surufatinib,AEs/SAEs were evaluated using NCI-CTCAE v5.0
Disease Control Rate(DCR) | 6 months after the last patient enrolled
  DCR was defined as the percentage of patients with complete response (CR), partial response (PR) and stable disease (SD) according to Response Evaluation Criteria in Solid Tumours (RECIST).
Overall survival (OS) | 6 months after the last patient enrolled
  OS was defined as the length of time from the administration of the first-dose until death from any cause.
  or lost of follow-up
Objective Response Rate (ORR) | 6 months after the last patient enrolled
  ORR was defined as the percentage of patients with complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST).

OTHER OUTCOMES:
QoL | 6 months after the last patient enrolled
  Using quality of life questionnaire (EORTC QLQ-C30) to collect the score. Scale range is 30~126, higher values are considered to be a better outcome.
Biomarkers | before the first dose
  Explore the correlation between curative effect and different biomarkers, such as EGFR mutation, FGFR etc.